CLINICAL TRIAL: NCT00308958
Title: Comparison of Airway Clearance Efficacy of Sine Wave and Triangular Wave High Frequency Chest Wall Oscillation (HFCWO) Devices in Patients With Cystic Fibrosis
Brief Title: Comparison of Airway Clearance Efficacy of Two High Frequency Chest Wall Oscillation (HFCWO) Devices in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0510M75246
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; chest physiotherapy; airway clearance; bronchiectasis
MeSH Terms: conditions — Cystic Fibrosis; Bronchiectasis

INTERVENTIONS:
Device: High frequency chest wall oscillator

SUMMARY:
Patients with cystic fibrosis (CF) must perform daily bronchial drainage therapy (BD) to keep their airways clear of secretions. Many different techniques are available to achieve this and there is currently no agreement as to which form of therapy is most effective. High frequency chest wall oscillation (HFCWO is used for this purpose by CF patients throughout the United States and abroad. To perform this therapy, the patient wears a vest which fits over the entire torso and is connected to an air compressor. The compressor generates oscillating air pulses that are transmitted to the lungs, thereby mobilizing secretions. The oscillations produced by the most commonly used device have a sinusoidal wave form (The Vest™ Airway Clearance System, Hill-Rom Inc, St Paul, MN). Previous studies indicate this form of therapy is as effective as more traditional and cumbersome forms of therapy. The design of the pulse generator has been recently modified so that the oscillations produced have a triangular wave form (Respitech Inc, MN). Studies done at the University of Minnesota found that the air flows induced in the airways can vary substantially depending on the wave form applied to the chest. At present, the impact of using a triangular wave form on mucus removal is unknown. The proposed study will compare mucous clearance using a device generating sine wave oscillations to a device generating triangular wave oscillations.

Hypothesis: Bronchial drainage using a triangular wave form of HFCWO will result in superior sputum production compared to HFCWO using a sine wave form.

Secondary Hypotheses:

Bronchial drainage using a triangular wave form of HFCWO may result in sputum with rheologic properties distinct from sputum produced while using sine wave HFCWO.

Bronchial drainage using a triangular wave form of HFCWO may result in superior post-therapy pulmonary function tests compared to pulmonary function tests obtained following therapy with sine wave HFCWO.

Subjects will perceive bronchial drainage using a triangular wave form of HFCWO as more comfortable than airway clearance using sine wave HFCWO.

DETAILED DESCRIPTION:
Participation in the study will be for 4 days. During initial subject recruitment, investigators will review inclusion and exclusion criteria with potential subjects. Upon enrollment, qualifying subjects will be asked to perform their last BD of the day at 8 PM on the day, but will be allowed to continue with the rest of their routine therapeutic regimen (including aerosols). They will be instructed to come on day 1 of the study at 8 AM. During this visit, they will complete a brief questionnaire and undergo an abbreviated physical exam, concentrating on chest findings. The questionnaire and exam will be used to confirm all subjects meet the study inclusion and exclusion criteria. The current therapeutic regimen being followed on day one of the study will be reviewed and the patient will be asked not to make any changes during the study period. Subjects will then perform pulse oximetry, spirometry, and lung volumes via body plethysmography. A sputum specimen will be collected for rheologic studies in a special container.

Once this is completed, the patient will perform a 30 minute BD session according to the first treatment of the randomly allocated sequence. The vest, or jacket, worn by the subject differs for the sine wave and triangular wave devices. Subjects will be blinded as to the type of system used at each session. Blinding will be accomplished by the patient wearing eye blinds of the type used commercially for assisting sleep. Investigators will assist the patient with putting on the HFCWO device. A large, lightweight poncho will then be placed over the patients head, thereby concealing the vest and attached equipment. The blinds will then be removed and the patient will subsequently put on a set of ear protectors used commercially for workers with noise exposure. This will prevent the patients from recognizing the difference in the sounds produced by the two devices. Only the respiratory therapist supervising the session will know of the treatment assignment. It is possible the subjects will be able to differentiate the two devices despite these measures to blind treatment. Subjects will use the vest devices provided by the investigators rather than bringing their vest devices from home. Prior to initiating the study, both devices will be tested, and adjusted as necessary, to ensure "dialed in" pressures and frequencies are accurately delivered.

During this session all the sputum produced will be collected in pre-weighed special containers and sealed for immediate processing. Patients will use their routine combination of aerosols in conjunction with the BD session. At the end of the 30 minute session the patient will be asked to produce a second sputum specimen which will be collected for rheologic studies in a special container.

After this is completed, pulmonary function measurements will be repeated. The patient will then undergo an abbreviated physical exam and complete a brief questionnaire (included in this application). The 8-item survey instrument focuses on adverse effects and comfort associated with use of the HFCWO device, primarily using a 5-point scale. Responses to the experience of using each device will be compared using standard statistical methodology.

The patient will be discharged after the measurements are completed and will be asked to return 3 days later for the second treatment in the allocated sequence. The patient will be asked to continue in the interim with their daily routines, trying not to make major changes in physical activity, environmental exposures or fluid intake. For the second treatment, the patient will be instructed again to perform BD at 8 PM on the evening before the return appointment.

On the second visit, subjects will undergo the same routine followed during the first visit.

Sputum Measurements

All sputum that the patient produces during a therapy session will be collected in pre-weighed specimen containers and sealed immediately. After the specimen is weighed ('raw wet weight'), the specimen will be centrifuged at 27,000 g for 15 minutes at 4oC and the supernatant will be carefully and completely discarded. This step eliminates any fluid coming from saliva that may have contaminated the specimen. The container with the sputum pellet will be weighed again ('wet weight') and left open in an oven with the temperature set at 150o F for 3 days to allow for complete desiccation. After this, the container will be weighed again to determine the sputum 'dry weight'. The 'raw wet weight' of the specimen collected at the end of the session for rheologic studies will be recorded and its dry weight will be calculated by extrapolation from the 'wet weight' and 'dry weight' obtained in the larger specimen. The addition of the weights for these two specimens will give the total sputum production for the session.

Pulmonary function testing

Patients will perform spirometry and lung volumes determination by body plethysmography at baseline and at the end of each BD session. At the same time, oxygen saturation will be determined by earlobe pulse oxymetry. Forced vital capacity (FVC) and Forced expiratory volume in 1 second (FEV1) will be obtained from the spirometry results; patients will perform single-breath nitrogen washout. All tests will be performed following the techniques which are already standard at the pediatric pulmonary laboratory and which follow the strict American Thoracic Society guidelines . All results will be expressed as the percent of predicted for age, gender and height.

Sputum Rheologic Properties The specimen collected at the end of each session will be weighed and frozen immediately at -70oC. The samples will be sent later to Dr. Bruce Rubin, Wake Forest University, Winston-Salem NC for further study.

E. Data Analysis.

Primary outcome: For each patient the sputum production during each treatment period will be determined by recording the total 'wet' sputum weights obtained during each treatment period. Sputum weights will be averaged for each treatment arm to obtain the mean 'wet' sputum productions for each treatment, and analyzed by analysis of variance for differences between the means. The sputum dry weights will be analyzed similarly.

Secondary outcomes: Percent change will be calculated for the FVC, FEV1, and Single-breath nitrogen washout seen in each patient during a given treatment period. The mean percent change will be calculated for each treatment and differences between these will be analyzed by analysis of variance. The same procedure will be followed for the rheologic measures.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CF established by sweat chloride > 60 mmol/L.
2. Age older than 18 years.
3. History of chronic daily sputum production.
4. Currently on a home therapeutic regimen that includes some form of BD performed at least 2 times daily that also includes concomitant use of an inhaled mucolytic and inhaled bronchodilator.
5. FVC and FEV1 > 40%-predicted, and with stable lung function (no greater than a 10% variation in lung function parameters over the preceding 4 months).
6. Evaluated at the University of Minnesota CF Center 3 or more times in the preceding 12 months.

Exclusion Criteria:

1. Hospitalization for CF pulmonary complications in the 2 months preceding enrollment.
2. Hemoptysis > 60 cc in a single episode in the 4 weeks preceding enrollment.
3. Chronic chest pain.
4. Participation in another clinical trial in the previous 30 days.
5. Use of intravenous antibiotics in the 2 months preceding enrollment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2006-02; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Average sputum production, as assessed by sputum wet and dry weights, during each treatment session.

SECONDARY OUTCOMES:
Change in pulmonary function parameters (Forced Vital Capacity and Forced Expiratory Volume in 1 second and Single-breath Nitrogen Washout) before and after therapy session for each of the treatment periods.
Sputum rheologic properties (adhesivity, cohesivity and viscoelastic parameters) for each treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Kempainen, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Kempainen RR, Williams CB, Hazelwood A, Rubin BK, Milla CE. Comparison of high-frequency chest wall oscillation with differing waveforms for airway clearance in cystic fibrosis. Chest. 2007 Oct;132(4):1227-32. doi: 10.1378/chest.07-1078. Epub 2007 Sep 21. PMID 17890465